CLINICAL TRIAL: NCT01167959
Title: Hypothalamic Morphology, Neuronal Activity and Systems Biology in Response to Food Intake in Obese Patients With Type 2 Diabetes Mellitus Compared to Obese and Lean Controls
Brief Title: Hypothalamic Function Before and After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Mirjam Anne Lips, drs, Leiden University Medical Center
Other Study IDs: P08-215
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Obesity; Diabetes
Keywords: Obesity; Diabetes; Bariatric surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood/Sera Adipose tissue biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- obesity diabetes, surgical and dietary
  Interventions: Procedure: Roux en Y gastric bypass and lap. gastric banding; Behavioral: Prodimed dietary intervention

INTERVENTIONS:
Procedure: Roux en Y gastric bypass and lap. gastric banding — Standard RYGB and LAGB procedures
Behavioral: Prodimed dietary intervention — 3 months of using the prodimed diet

SUMMARY:
The purpose of this study is to determine the effect of gastric banding or gastric bypass on hypothalamic morphology and function, gut hormones and systems biology in obese subjects with and without type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35-65 years;
* BMI > 40 kg/m2;
* BMI > 35 and <40 kg/m2 with co-morbidity, which is expected to improve after surgically-induced weight loss;
* A history of longstanding obesity (>5 years);
* Proven failed attempts to lose weight in a conventional way, or primarily successful weight loss with eventual weight regain;
* Intention to adhere to a postoperative follow-up programme.

Exclusion Criteria:

* BMI> 50 or body weight > 150 kg (because it is impossible to safely put people above this weight on a standard table for MRI);
* Subjects with disease related obesity, i.e. Cushing or medication related obesity;
* Use of medication known to affect glucose or lipid metabolism (i.e. prednisone)
* Monogenetic diabetes: MODY, Mitochondrial diabetes;
* LADA (adult-onset latent autoimmune diabetes); detected by c-peptide measurement on screening.
* Impaired renal function (serum creatinine > 176 μmol/L);
* Leg ulcers, gangrene.
* Any genetic or psychiatric disease (e.g. fragile X syndrome, major depression) affecting the brain
* Any significant chronic disease
* Renal or hepatic disease
* Pregnancy
* Recent weight changes or attempts to loose weight (> 3 kg weight gain or loss, within the last 3 months)
* Aerobic exercise more that 3 times 60 minutes a week
* Alcohol consumption of more than 28 units per week at present or in the past
* Recent blood donation (within the last 2 months)
* Recent participation in other research projects (within the last 3 months), participation in 2 or more projects in one year
* Contra-indications to operative procedures as regular in bariatric surgery
* Contra-indications to MRI scanning

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese (type 2 diabetic or not) population from primary care (dietary intervention) and hospital setting (bariatric surgery)
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Changes in gut hormones | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hanno Pijl, MD Phd Proff, Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

REFERENCES:
- [Derived] Maessen DE, Hanssen NM, Lips MA, Scheijen JL, Willems van Dijk K, Pijl H, Stehouwer CD, Schalkwijk CG. Energy restriction and Roux-en-Y gastric bypass reduce postprandial alpha-dicarbonyl stress in obese women with type 2 diabetes. Diabetologia. 2016 Sep;59(9):2013-7. doi: 10.1007/s00125-016-4009-1. Epub 2016 Jun 16. PMID 27312699
- [Derived] Lips MA, Van Klinken JB, van Harmelen V, Dharuri HK, 't Hoen PA, Laros JF, van Ommen GJ, Janssen IM, Van Ramshorst B, Van Wagensveld BA, Swank DJ, Van Dielen F, Dane A, Harms A, Vreeken R, Hankemeier T, Smit JW, Pijl H, Willems van Dijk K. Roux-en-Y gastric bypass surgery, but not calorie restriction, reduces plasma branched-chain amino acids in obese women independent of weight loss or the presence of type 2 diabetes. Diabetes Care. 2014 Dec;37(12):3150-6. doi: 10.2337/dc14-0195. Epub 2014 Oct 14. PMID 25315204
- [Derived] Lips MA, Wijngaarden MA, van der Grond J, van Buchem MA, de Groot GH, Rombouts SA, Pijl H, Veer IM. Resting-state functional connectivity of brain regions involved in cognitive control, motivation, and reward is enhanced in obese females. Am J Clin Nutr. 2014 Aug;100(2):524-31. doi: 10.3945/ajcn.113.080671. Epub 2014 Jun 25. PMID 24965310
- [Derived] Lips MA, Pijl H, van Klinken JB, de Groot GH, Janssen IM, Van Ramshorst B, Van Wagensveld BA, Swank DJ, Van Dielen F, Smit JW. Roux-en-Y gastric bypass and calorie restriction induce comparable time-dependent effects on thyroid hormone function tests in obese female subjects. Eur J Endocrinol. 2013 Aug 28;169(3):339-47. doi: 10.1530/EJE-13-0339. Print 2013 Sep. PMID 23811187